CLINICAL TRIAL: NCT01673971
Title: Optical Tomographic Imaging of Infantile Hemangiomas
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Maria Garzon, Professor of Clinical Dermatology and Clinical Pediatrics, Columbia University
Other Study IDs: AAAJ1201
Record Dates: First submitted 2012-08-24; First posted 2012-08-28 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Infantile Hemangioma
Keywords: hemangioma
MeSH Terms: conditions — Hemangioma, Capillary; Hemangioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Natural History
- Treatment

SUMMARY:
The investigators hypothesize that there are differences between infantile hemangiomas (IH) during the proliferating and involuting phases and in response to medical treatment that can be detected by optical tomography of these hemangiomas.

DETAILED DESCRIPTION:
Infantile hemangiomas (IH) are common vascular growths that frequently arise in infants. The clinical presentation is variable, and some hemangiomas have the potential to cause disfiguring and even lifethreatening complications. While there is no FDA approved treatment for IH, certain medications have been shown to be effective in shrinking the growths. Unfortunately, there is no objective tool to monitor IH or to guide treatment. Such a tool would improve the management of these patients. A new handheld wireless device uses diffuse optical imaging (DOI) technology to measure blood flow characteristics.

The device has been used in studies to assess patients with breast cancer. Optical tomography has also been increasingly used to assess neurological function and pathology in newborn infants.

The goal of the investigators' study is to assess the utility of DOI for characterizing and monitoring IH. Fifteen IH will be assessed at three points in time as part of this study, comprising two groups: 'Natural History' and 'Treatment'. DOI measurements will be correlated with clinical findings and existing ultrasound measurements of the IH.

ELIGIBILITY:
For the 'Natural History' Cohort, the following inclusion and exclusion criteria apply:

INCLUSION CRITERIA:

* Infants with IH who present to our practices within the first 2 months of life.
* IH of size > 2 cm in diameter
* IH located on area of skin that is accessible to contact by 4x2cm probe. Examples include the lateral face, forehead, scalp, trunk and areas of the extremities not overlying joints.

Infants with IH that do not necessitate either medical or surgical intervention at time of presentation.

EXCLUSION CRITERIA:

* IH of size <2 cm in diameter
* Complicated IH requiring medical or surgical intervention
* IH located within 2 cm of the eye

For the 'Treatment' Cohort, the following inclusion and exclusion criteria apply:

INCLUSION CRITERIA:

* Infants with IH who present to our practices within the first 2 months of life.
* IH of size >2 cm in diameter
* IH located on area of skin that is accessible to contact by 4x2cm probe. Examples include the lateral face, forehead,scalp, trunk and areas of the extremities not overlying joints.
* IH that necessitate medical intervention with either oral or topical betablockers.

EXCLUSION CRITERIA:

* IH <2 cm in size
* Complicated IH requiring surgical intervention
* IH located within 2 cm of the eye

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All subjects will be recruited verbally from the pediatric dermatology faculty practices, clinics and inpatient services at CUMC/NYP (MSCHONY). In accordance with CUMC policy, researchers will not approach a patient for recruitment until that patient has been informed of the study by their treating physician who has ascertained the patient's willingness to discuss the study with the investigators.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-05; Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Difference in absolute total hemoglobin concentration ([THb]) of hemangioma and normal skin. | Up to 2 years
  Measurements of absolute total hemoglobin concentration ([THb]) of hemangioma and normal skin are obtained using a diffuse optical imaging device and are compared at different time points.
Difference in tissue oxygen saturation (StO2) of hemangioma and normal skin. | Up to 2 years
  Measurements of tissue oxygen saturation (StO2) of hemangioma and normal skin are obtained using a diffuse optical imaging device and are compared at different time points.

SECONDARY OUTCOMES:
Difference in absolute total hemoglobin concentration ([THb]) of hemangioma at different time points. | Up to 2 years
  Measurements of absolute total hemoglobin concentration ([THb]) of the hemangioma are obtained at different time points and compared.
Difference in tissue oxygen saturation (StO2) of the hemangioma at different time points. | Up to 2 years
  Measurements of tissue oxygen saturation (StO2) of the hemangioma are obtained at different time points and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Garzon, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center / Department of Dermatology, New York, New York, United States